CLINICAL TRIAL: NCT01055899
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety and Tolerability of Subcutaneously Administered REGN88 in Subjects With Rheumatoid Arthritis Receiving Concomitant Methotrexate
Brief Title: Safety Study of a Single Dose of REGN88(SAR153191)in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6R88-RA-0801
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 (Experimental): First dose of SC REGN88
  Interventions: Biological: REGN88
- Dose 2 (Experimental): Second dose of SC REGN88
  Interventions: Biological: REGN88
- Dose 3 (Experimental): Third dose of SC REGN88
  Interventions: Biological: REGN88

INTERVENTIONS:
Biological: REGN88 — Single SC Dose
  Arms: Dose 1
Biological: REGN88 — Single SC Dose
  Arms: Dose 2
Biological: REGN88 — Single SC Dose
  Arms: Dose 3

SUMMARY:
This study will test the safety and tolerability (how the body reacts to the drug) of REGN88 and placebo (an inactive substance that contains no medicine) in patients with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blind, placebo-controlled, single dose escalation study of the safety and tolerability of subcutaneously administered REGN88 in rheumatoid arthritis patients who are receiving concomitant methotrexate.

Three (3) sequential dose cohorts of 5 subjects (4:1 active: placebo) will be dosed SC with REGN88 or placebo. Subjects who complete the study will participate in 14 study visits over 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Subjects must weigh > 50 kg and < 100 kg
3. Diagnosis of Rheumatoid Arthritis (RA) as defined by the 1987 revised American College of Rheumatology (ACR) criteria with disease duration of no less than 6 months and ACR class I-III
4. For women of childbearing potential, a negative serum pregnancy test at the Screening Visit (Visit 1) and a negative urine pregnancy test at Day -1
5. For men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner[s] become pregnant) during the full course of the study.

Exclusion Criteria:

1. A history of Listeriosis or active tuberculosis (TB)
2. Persistent chronic or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the Screening Visit
3. History of prior articular or prosthetic joint infection
4. History of a hypersensitivity reaction, other than localized injection site reaction (ISR), to any biological molecule
5. Significant concomitant illness such as, but not limited to cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease that would adversely affect the subject's participation in this study
6. Received administration of any live (attenuated) vaccine within 3 months prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of a single dose of subcutaneously administered REGN88 in subjects with rheumatoid arthritis who are receiving concomitant treatment with methotrexate | 113 Days

SECONDARY OUTCOMES:
To assess the PK profile of a single subcutaneous (SC) dose of REGN88, and the immunogenicity of a single SC dose of REGN88 | 113 days

CONTACTS AND LOCATIONS:
Overall Officials: Allen Radin, M.D., Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Duncansville, Pennsylvania
  - Dallas, Texas